CLINICAL TRIAL: NCT03667768
Title: Atraumatic Restorative Treatment Sealants in First Permanent Molars: a Bi-center Split-mouth Clinical Trial
Brief Title: Atraumatic Restorative Treatment Sealants in First Permanent Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Academic Centre for Dentistry in Amsterdam (Other); Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Daniela Hesse, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: USP-SaoPaulo
Record Dates: First submitted 2018-08-21; First posted 2018-09-12 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Caries, Dental
Keywords: Dentition, Permanent; Glass Ionomer Cements
MeSH Terms: conditions — Dental Caries | interventions — Toothbrushing

STUDY DESIGN:
Intervention Model Description: Split-mouth design
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glass ionomer sealant (Experimental): Two hand-mixed glass ionomer cements (GICs) available in the dental market were used, and they were mixed according to the manufacturer's instructions (powder/liquid ratio 1:1). The molars were cleaned with a toothbrush and wet cotton wool pellets. Isolation was performed with cotton wool rolls and the occlusal surface was conditioned with GIC liquid (20s), rinsed with wet cotton wool pellets and dried with dry cotton wool pellets. GIC was placed on the occlusal surface and pressed into the pits and fissures using the press-finger technique. The excess of material was removed and the occlusion checked and adjusted. Sealant was protected with a new layer of petroleum jelly and the children were instructed not to eat for at least one hour. Children received instructions on how to brush their teeth (1,000-ppm fluoridated dentifrice), as well as advices regarding diet and information about dental caries was given by a dental assistant and those instructions were repeated every 6 months.
  Interventions: Procedure: Glass ionomer sealant
- Non-sealant (toothbrushing) (Other): No sealant was performed. Children received instructions on how to brush their teeth (1,000-ppm fluoridated dentifrice), as well as advices regarding diet and information about dental caries was given by a dental assistant and those instructions were repeated every 6 months.
  Interventions: Behavioral: Non-sealant (toothbrushing)

INTERVENTIONS:
Procedure: Glass ionomer sealant
  Arms: Glass ionomer sealant
Behavioral: Non-sealant (toothbrushing)
  Arms: Non-sealant (toothbrushing)

SUMMARY:
The aim of this bi-center study was to evaluate the retention and caries-preventive effect of Atraumatioc Restorative Treatment (ART) sealants, using two glass ionomer cement (GIC) versus non-sealant on first permanent molars of schoolchildren. The null hypothesis is that there is no difference in the retention rates of the two GIC, as well as in caries prevention between sealants application and non-sealant. Four hundred and thirty-seven 6-to-8-year-old schoolchildren were selected in two cities in Brazil. They were randomly divided into two groups, according to the GIC used (Fuji IX or Maxxion). All children had their four first permanent molars included in the research and two molars were sealed with a GIC, while the other two molars remained unsealed. Clinical evaluations were performed up to 36 months by one independent examiner at each city.

ELIGIBILITY:
Inclusion Criteria:

* patients presenting the four first permanent molars without gingival tissue covering the occlusal surface and without clinically detectable dentine caries lesion, assessed as scores 0, 1 and 2 of ICDAS criteria [Ismail AI, Sohn W, Tellez M, et al (2007) The International Caries Detection and Assessment System (ICDAS): An integrated system for measuring dental caries: Methods. Community Dent Oral Epidemiol 35:170-178 ].

Exclusion Criteria:

* patients presenting any physical and/or medical health issues and having non-cooperative behavior.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 437 (Actual)
Dates: Start 2010-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Changes in glass ionomer selants retention | 3, 6, 12, 18, 24 and 36 months
  The sealants retention was evaluated clinically using the criteria: 0) fully present sealant; 1) partially present sealant and 2) absent sealant [Oba AA, Dülgergil T, Sönmez IŞ, Doǧan S (2009) Comparison of Caries Prevention With Glass Ionomer and Composite Resin Fissure Sealants. J Formos Med Assoc 108:844-848]. Scores 0 and 1 were considered "success," whereas score 2 was considered "failure."

SECONDARY OUTCOMES:
Changes in caries status of first permanent molars | 3, 6, 12, 18, 24 and 36 months
  The examiners evaluated the presence of caries according to ICDAS [Ismail AI, Sohn W, Tellez M, et al (2007) The International Caries Detection and Assessment System (ICDAS): An integrated system for measuring dental caries: Methods. Community Dent Oral Epidemiol 35:170-178] and caries activity according to Nyvad criteria [Nyvad B, Machiulskiene V, Baelum V (1999) Reliability of a New Caries Diagnostic System Differentiating between Active and Inactive Caries Lesions. Caries Res 33:252-260].
  ICDAS codes 0 to 4 indicated success, while codes 5 and 6 were considered failures.
Comparison between the development of caries in dentine(measured using ICDAS score system) of first permanent molars between the two cities | 3, 6, 12, 18, 24 months
  The examiners evaluated the presence of caries according to ICDAS [Ismail AI, Sohn W, Tellez M, et al (2007) The International Caries Detection and Assessment System (ICDAS): An integrated system for measuring dental caries: Methods. Community Dent Oral Epidemiol 35:170-178] and caries activity according to Nyvad criteria [Nyvad B, Machiulskiene V, Baelum V (1999) Reliability of a New Caries Diagnostic System Differentiating between Active and Inactive Caries Lesions. Caries Res 33:252-260]. The comparison between the 2 cities was performed in order to verify if demographic/ population characteristics could interfere in the treatments. ICDAS codes 0 to 4 indicated success, while codes 5 and 6 were considered failures.

IPD SHARING:
Plan to Share IPD: No